CLINICAL TRIAL: NCT02061020
Title: Pilot Study of the Relationship Between Dose-concentration-effect of Delta-9-tetrahydrocannabinol and the Ability to Drive in Chronic or Occasional Cannabis Users
Brief Title: Study of the Relationship Between Dose-concentration-effect of Delta-9-tetrahydrocannabinol (THC) and the Ability to Drive in Chronic or Occasional Cannabis Users
Acronym: VIGICANN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AOR12144 / P111114; 2013-A00245-40 (Other: IDRCB)
Record Dates: First submitted 2013-12-18; First posted 2014-02-12 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-05

CONDITIONS: Occasional (1-2 Joints Per Week) and Chronic (1-2 Joints Per Day) Cannabis Users
Keywords: delta-9-tetrahydrocannabinol, volunteers, cannabis users
MeSH Terms: interventions — nabiximols; Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sequence 1 (Experimental): 1. THC containing cigarettes 10mg
  2. THC containing cigarettes 30mg
  3. Placebo
  Interventions: Drug: Cannabis (THC) in cigarettes of 30mg, 10mg and placebo
- Sequence 2 (Experimental): 1. THC containing cigarettes 30mg
  2. Placebo
  3. THC containing cigarettes 10mg
  Interventions: Drug: Cannabis (THC) in cigarettes of 30mg, 10mg and placebo
- Sequence 3 (Experimental): 1. Placebo
  2. THC containing cigarettes 10mg
  3. THC containing cigarettes 30mg
  Interventions: Drug: Cannabis (THC) in cigarettes of 30mg, 10mg and placebo

INTERVENTIONS:
Drug: Cannabis (THC) in cigarettes of 30mg, 10mg and placebo — Smoked THC containing cigarettes. Randomly allocated dosage 30mg, 10mg et placebo.
  Both chronic and occasional cannabis consuming volunteers will be allocated to smoking a cigarette containing (1) no THC (placebo), (2) a joint containing 1% THC (10 mg THC, i.e. low-dose) and (3) a joint containing 3% (30 mg THC) mixed with 1 g tobacco.
  Each cigarette will be followed by 24 hours testing in laboratory conditions. Each period is separated by 7 days (3 testing periods over 3 weeks). Each volunteer will undergo performance testing (driving simulator and PVT) before administration of the substance (T0).
  Blood samples and repeat performance testing will be carried out at 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours and 24 hours.

SUMMARY:
Study of the effects of smoked cannabis consumption on performance on a driving simulator and reaction time. The study aims to explore the relationship between concentrations of cannabis in the blood, driving performance and reaction time.

DETAILED DESCRIPTION:
This study will examine:

* The relationship between THC blood levels and driving performance measured on a York Driving simulator
* The relationship between THC blood levels and reaction times as measured on the psychomotor vigilance test (PVT)
* the pharmacokinetics of THC in occasional and chronic cannabis consumers
* Determine the minimum blood concentration level of THC and 11-OH-THC, below which no effect of cannabis is observed
* Determine whether the polymorphism of CYP2C9 (* 3) is associated with the AUC, Cmax, and higher THC T1/2
* Determine if the polymorphism of CYP2C9 (* 3) is associated with different pharmacodynamic effects at a given THC level on performance measured by driving simulation

ELIGIBILITY:
Inclusion criteria:

* Healthy volunteer of male gender from 18 to 25 years
* Normal medical examination
* Driving license owner
* BMI between 18.5 and 25
* moderate tobacco consumption
* moderate consumption of coffee, tea, cola (≤ 225mg caffeine per day)
* Cannabis user for at least 1 year
* Occasional (1-2 joints per week) or chronic (1-2 joints per day) cannabis consumers
* Availability during the study
* Signed consent

Exclusion criteria:

* Participation in another clinical study
* Having taken any psychotropic medication in the past one month
* Having taken any narcotic (alcohol, psychotropic drugs, other narcotics) other than THC in the past 3 days (negative urinary test at inclusion)
* Alcohol blood level positive at inclusion
* Excessive alcohol consumption (AUDIT score > 7)
* Dependence, present or past, to any psychotropic product (alcohol, psychoactive drugs, other narcotic)
* Depression
* Sleep disorders
* Any psychiatric history, including psychosis
* Deprived of their liberty by judicial or administrative decision
* Lack of medical insurance
* Professional use of motorized vehicles

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2014-01; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Ability to drive a motor vehicle measured using a driving simulator | 0h, 1h, 2h, 4h, 6h, 8h, 12h and 24 h
  The association between THC blood concentrations and driving performances as measured by deviations from the centre of the road and variations of speed at 0h, 1h, 2h, 4h, 6h, 8h, 12h and 24 h after smoking.

SECONDARY OUTCOMES:
Psychomotor Vigilance Test (PVT) measures | 0h, 1h, 2h, 4h, 6h, 8h, 12h et 24h
  The association between THC blood concentration and impaired reaction time on PVT measured sequentially over 24 hours
THC pharmacokinetics of occasional and chronic users over 24 hours | 24 hours
  THC pharmacokinetics parameters (AUC, T1/2, CMAX) of occasional and chronic users over 24 hours will be modelled using a population nonlinear mixed approach.
24 hoursTHC pharmacokinetics (AUC, T1 / 2, CMAX) and its relationships with genotype CYP2C9 * 3 | 24 hours
  24 hoursTHC pharmacokinetics (AUC, T1 / 2, CMAX) and its relationships with genotype CYP2C9 * 3

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hartley, MD, Principal Investigator — Sleep Disorders Unit - Raymond Poincaré Hospital
Locations (1):
- Raymond Poincare Hospital, Garches, France

REFERENCES:
- [Derived] Hartley S, Simon N, Cardozo B, Larabi IA, Alvarez JC. Can inhaled cannabis users accurately evaluate impaired driving ability? A randomized controlled trial. Front Public Health. 2023 Nov 22;11:1234765. doi: 10.3389/fpubh.2023.1234765. eCollection 2023. PMID 38074719
- [Derived] Alvarez JC, Hartley S, Etting I, Ribot M, Derridj-Ait-Younes N, Verstuyft C, Larabi IA, Simon N. Population pharmacokinetic model of blood THC and its metabolites in chronic and occasional cannabis users and relationship with on-site oral fluid testing. Br J Clin Pharmacol. 2021 Aug;87(8):3139-3149. doi: 10.1111/bcp.14724. Epub 2021 Jan 12. PMID 33386756
- [Derived] Hartley S, Simon N, Larabi A, Vaugier I, Barbot F, Quera-Salva MA, Alvarez JC. Effect of Smoked Cannabis on Vigilance and Accident Risk Using Simulated Driving in Occasional and Chronic Users and the Pharmacokinetic-Pharmacodynamic Relationship. Clin Chem. 2019 May;65(5):684-693. doi: 10.1373/clinchem.2018.299727. Epub 2019 Mar 14. PMID 30872375